CLINICAL TRIAL: NCT00746577
Title: Organizational Factors Influencing Practice Improvement in Community Based
Brief Title: Organizational Factors Influencing Practice Improvement in Community Based Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Richmond Behavioral Health Authority (RBHA) (Unknown); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01DA022081 (NIH); R01DA022081 (NIH)
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2011-10

CONDITIONS: Quality of Treatment Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Organizational change to improve the implementation of evidence-based practices. — Some sites will receive assistance with the creation and implementation of an organizational development plan.

SUMMARY:
Purpose of the Study:

The Richmond Behavioral Health Authority's Substance Abuse Services Division and Virginia Commonwealth University's Institute for Drug and Alcohol Studies are working on an important research study to improve the quality of substance use disorder treatment services offered by RBHA and its contracted services providers. Specifically, this preliminary research will provide the information needed to conduct a planned series of program-specific interventions, designed to increase the adoption of evidence-based practices (EBPs) within specific programs. A major goal of the study is to better understand what factors influence the adoption of EBPs, and what adoption strategies work best for which types of staff, which types of programs, and under what conditions.

Description of Staff Involvement:

In this study, staff will be asked to complete questionnaires about themselves, their workplaces, and their perceptions about the services their organization provides. Some of these questionnaires will be given to staff when they first enter the study, and others may be given to staff before and about 9 months after a 3-day Practice Improvement Workshop (please note that each agency may or may not be selected to complete the workshop).

Description of Client Involvement:

Clients at each participating site will be asked to complete a brief survey about the services they receive at that site. This survey will occur at the initial timepoint, and at several later timepoints. This survey is confidential and anonymous.

ELIGIBILITY:
Inclusion Criteria:

* Substance abuse staff members (who work with adults) working at Richmond Behavioral Health Authority (RBHA) and its contracted providers
* Clients seen at RBHA and its contracted providers during specific periods, who are at least 18 years of age

Exclusion Criteria:

* Being under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 910 (Actual)
Dates: Start 2008-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Survey | Pre and post intervention

SECONDARY OUTCOMES:
Data from database of client information | Pre and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: James C May, PhD, Principal Investigator — Richmond Behavioral Health Authority (RBHA)
Locations (1):
- Richmond Behavioral Health Authority, Richmond, Virginia, United States